CLINICAL TRIAL: NCT06696859
Title: Patterns of Antibiotics Resistance Among Respiratory ICU Patients
Brief Title: Patterns of Antibiotics Resistance
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Safaa Saber Aly, Resident at Chest Diseases Department, Sohag University
Other Study IDs: Soh-Med-15-10_14MS
Record Dates: First submitted 2024-11-08; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Antibiotics Resistance
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antibiotics — Bacterial culture (sputum ,blood and pleural fluid) Antibiotics sensitivity tests

SUMMARY:
Antibiotics resistance has become a global health challenge especially in third world countries. The main causes of antibiotics resistance are the improper use or overuse of antibiotics, the lack of skilled public health workers and poor hygiene standards. Resistance to antibiotics reduces the effectiveness of these treatments and has a negative impact on hospital systems especially in intensive care settings.

Medical intensive care unit (MICU) is commonly known as a "hotbed of infections" in high-risk healthcare environments ICU patients are especially prone to infections because of the various invasive procedures they undergo,including vascular access, mechanical ventilation, and intubation.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be admitted at respiratory ICU with respiratory infection who have been treated with antibiotics and patients in whom adequate respiratory specimen is obtained will be included in the study

Exclusion Criteria:

* Patients who are HIV positive, who can't provide adequate respiratory specimen, patients who are not on antibiotics and patients who die within 48 hours after admission

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients will be admitted at respiratory ICU with respiratory infection who have been treated with antibiotics and patients in whom adequate respiratory specimen
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Patterns of Antibiotics Resistance | 6months to 1 year
  Number of resistance to antibiotics among ICU patients